CLINICAL TRIAL: NCT01607073
Title: Verapamil as Adjunctive Seizure Therapy for Children and Young Adults With Dravet Syndrome
Brief Title: Verapamil as Therapy for Children and Young Adults With Dravet Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gillette Children's Specialty Healthcare (Other)
Collaborators: Mayo Clinic (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IND 113666
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Dravet Syndrome
Keywords: Dravet; seizures; verapamil
MeSH Terms: conditions — Epilepsies, Myoclonic; Seizures | interventions — Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open label adjunctive add on (Other): open label adjunctive add on of verapamil to existing medications. dosing begins at 1 mg/kg/d and increases weekly to target of 4 mg/kg/d in divided doses (three times/day)
  Interventions: Drug: Verapamil

INTERVENTIONS:
Drug: Verapamil — Verapamil will be prepared as a solution. A 50mg/ml oral suspension may be made with immediate release tablets and either a 1:1 mixture of Ora-Sweet and Ora-Plus or a 1:1 mixture of Ora-Sweet SF and Ora-Plus will be used.
  Children will start on a 4 weeks titration period:
  Week 1: 1mg/kg/day divided BID Week 2: 2mg/kg/day divided BID or TID Week 3: 3mg/kg/day divided BID or TID Week 4: 4mg/kg/day divided TID
  In event of adverse events, and in consultation with the family and treating physician, the dosage may be decreased to 2mg/kg/day and remain at that dose for the remainder of the study.
  Other Names: Calan; Covera; Isoptin; Verelan

SUMMARY:
This study will assess how well the drug verapamil can improve control of seizures and dysautonomia symptoms in children and young adults diagnosed with Dravet syndrome. The safety of verapamil when given with all concomitant medications will also be assessed.

DETAILED DESCRIPTION:
Dravet syndrome (DS) is a devastating form of pediatric seizure disorder (epilepsy), often related to abnormalities of one of the genes that controls sodium channel function in the brain (SCN1A). Most children with DS experience continued seizures even with optimal treatment of currently available anti-seizure therapies [1]. Many of these seizures are prolonged, and can be life threatening.

This pilot study will assess the efficacy of verapamil in improving control of seizures in children and young adults DS. This will be done by adding verapamil as open label adjunctive therapy to medications already being given. Investigators will assess the effect of verapamil therapy on seizure control and on signs of autonomic dysfunction observable to the parents/guardians. Signs of autonomic function include body temperature regulation, sweating, heart rate, pupil size, and flushing of the skin. Iannetti, et al reported treating 2 children with clinical DS (one with an SCN1A mutation) with verapamil as adjunctive therapy [2]. Both children had a positive clinical response persisting for a number of months. No adverse effects were noted. We have treated an additional 4 children with DS with verapamil. There have been no significant adverse effects; 3 of 4 have experienced improved seizure control for months also.

Verapamil has been shown to affect autonomic tone in patients with cardiac disorders (eg. high blood pressure, heart attack). It alters the balance between parts of the autonomic nervous system's function (called sympathetic and parasympathetic function) with a shift toward decreased sympathetic tone and increased parasympathetic (vagus nerve) tone [8, 9, 10]. Verapamil is used as an effective agent to treat certain types of autonomic headaches in both adults and children. In cluster headaches, autonomic symptoms (tearing, nasal congestion, facial sweating, papillary constriction) are prominent; verapamil is an accepted treatment [11, 12].

Intense emotion triggers seizures in a subset of children with DS. Modulation of autonomic function is likely an integral part of seizure threshold in those so affected. Children with DS have a higher rate of signs of abnormal autonomic function than do controls [13]. Cardiac autonomic control is also altered in these children, with a shift in the balance between sympathetic (relatively overactive) and parasympathetic (relatively less active) tone [14]. Similar findings have been identified in adults with intractable epilepsy and children with partial epilepsy [15, 16, 17]. Verapamil's action in stabilizing the balance of sympathetic and parasympathetic tone may play a role altering autonomic tone abnormalities in children with DS as well. This may be a part of the mechanism that leads to improved seizure control.

Verapamil has been in clinical use for ~ 25 years. The FDA has granted an Investigational New Drug approval for use of this medication in this population of children and young adults. Investigators propose to add it to the patient's existing medications, and evaluate potential improvement in seizure control. Potential side effects will be screened. Investigators will monitor liver function with blood tests as well as concentrations of anti-seizure medications. Verapamil and nor-verapamil levels will be assessed twice also. Testing of heart rhythm (EKG) will be done before the study starts and twice more during the study.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 25 years old
* Onset of seizures in first year of life
* seizure type usually generalized tonic-clonic, clonic, or hemiclonic, often prolonged (>10 minutes)
* myoclonic jerks/myoclonic seizures
* history of normal development at seizure onset with subsequent developmental delay or regression which occurs after seizure onset
* presence of documented abnormality on the SCN1A gene
* medically intractable epilepsy: must have been on at least 2 prior antiepileptic medications without adequate control of epilepsy
* subject is capable of giving informed consent (or assent if possible) or has an acceptable surrogate capable of giving informed consent on the subject's behalf

Exclusion Criteria:

* use of clonidine, propranolol, carbamazepine, oxcarbazine, stiripentol, lamotrigine, or cyclosporine
* Abnormalities of cardiac conduction or rhythm (excluding sinus arrhythmia) on screening EKG
* significant use of grapefruit juice
* ketogenic diet
* pregnancy

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly S Wical, MD, Principal Investigator — Gillette Children's Specialty Healthcare
Locations (4):
- United States (4):
  - Children's Memorial Hospital, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Mary Hitchcock Memorial Hospital, Lebanon, New Hampshire

REFERENCES:
- [Background] Skluzacek JV, Watts KP, Parsy O, Wical B, Camfield P. Dravet syndrome and parent associations: the IDEA League experience with comorbid conditions, mortality, management, adaptation, and grief. Epilepsia. 2011 Apr;52 Suppl 2:95-101. doi: 10.1111/j.1528-1167.2011.03012.x. PMID 21463290
- [Background] Delogu AB, Spinelli A, Battaglia D, Dravet C, De Nisco A, Saracino A, Romagnoli C, Lanza GA, Crea F. Electrical and autonomic cardiac function in patients with Dravet syndrome. Epilepsia. 2011 Apr;52 Suppl 2:55-8. doi: 10.1111/j.1528-1167.2011.03003.x. PMID 21463281
- [Background] Iannetti P, Parisi P, Spalice A, Ruggieri M, Zara F. Addition of verapamil in the treatment of severe myoclonic epilepsy in infancy. Epilepsy Res. 2009 Jul;85(1):89-95. doi: 10.1016/j.eplepsyres.2009.02.014. Epub 2009 Mar 20. PMID 19303743
- [Background] Schwartz JB, Keefe DL, Kirsten E, Kates RE, Harrison DC. Prolongation of verapamil elimination kinetics during chronic oral administration. Am Heart J. 1982 Aug;104(2 Pt 1):198-203. doi: 10.1016/0002-8703(82)90192-2. PMID 7102502
- [Background] Flynn JT, Pasko DA. Calcium channel blockers: pharmacology and place in therapy of pediatric hypertension. Pediatr Nephrol. 2000 Dec;15(3-4):302-16. doi: 10.1007/s004670000480. PMID 11149130
- [Background] Porter CJ, Garson A Jr, Gillette PC. Verapamil: an effective calcium blocking agent for pediatric patients. Pediatrics. 1983 May;71(5):748-55. PMID 6340050
- [Background] Sapire DW, O'Riordan AC, Black IF. Safety and efficacy of short- and long-term verapamil therapy in children with tachycardia. Am J Cardiol. 1981 Dec;48(6):1091-7. doi: 10.1016/0002-9149(81)90325-8. No abstract available. PMID 6795914
- [Background] Lefrandt JD, Heitmann J, Sevre K, Castellano M, Hausberg M, Fallon M, Fluckiger L, Urbigkeit A, Rostrup M, Agabiti-Rosei E, Rahn KH, Murphy M, Zannad F, de Kam PJ, van Roon AM, Smit AJ. The effects of dihydropyridine and phenylalkylamine calcium antagonist classes on autonomic function in hypertension: the VAMPHYRE study. Am J Hypertens. 2001 Nov;14(11 Pt 1):1083-9. doi: 10.1016/s0895-7061(01)02218-x. PMID 11724204
- [Background] Petretta M, Canonico V, Madrid A, Mickiewicz M, Spinelli L, Marciano F, Vetrano A, Signorini A, Bonaduce D. Comparison of verapamil versus felodipine on heart rate variability in hypertensive patients. J Hypertens. 1999 May;17(5):707-13. doi: 10.1097/00004872-199917050-00016. PMID 10403616
- [Background] Forslund L, Bjorkander I, Ericson M, Held C, Kahan T, Rehnqvist N, Hjemdahl P. Prognostic implications of autonomic function assessed by analyses of catecholamines and heart rate variability in stable angina pectoris. Heart. 2002 May;87(5):415-22. doi: 10.1136/heart.87.5.415. PMID 11997407
- [Background] May A, Leone M, Afra J, Linde M, Sandor PS, Evers S, Goadsby PJ; EFNS Task Force. EFNS guidelines on the treatment of cluster headache and other trigeminal-autonomic cephalalgias. Eur J Neurol. 2006 Oct;13(10):1066-77. doi: 10.1111/j.1468-1331.2006.01566.x. PMID 16987158
- [Background] Lampl C. Childhood-onset cluster headache. Pediatr Neurol. 2002 Aug;27(2):138-40. doi: 10.1016/s0887-8994(02)00406-x. PMID 12213616
- [Background] Mukherjee S, Tripathi M, Chandra PS, Yadav R, Choudhary N, Sagar R, Bhore R, Pandey RM, Deepak KK. Cardiovascular autonomic functions in well-controlled and intractable partial epilepsies. Epilepsy Res. 2009 Aug;85(2-3):261-9. doi: 10.1016/j.eplepsyres.2009.03.021. Epub 2009 May 5. PMID 19409754
- [Background] Ferri R, Curzi-Dascalova L, Arzimanoglou A, Bourgeois M, Beaud C, Nunes ML, Elia M, Musumeci SA, Tripodi M. Heart rate variability during sleep in children with partial epilepsy. J Sleep Res. 2002 Jun;11(2):153-60. doi: 10.1046/j.1365-2869.2002.00283.x. PMID 12028480
- [Background] Yang TF, Wong TT, Chang KP, Kwan SY, Kuo WY, Lee YC, Kuo TB. Power spectrum analysis of heart rate variability in children with epilepsy. Childs Nerv Syst. 2001 Oct;17(10):602-6. doi: 10.1007/s003810100505. PMID 11685522
- [Background] Chiron C, Marchand MC, Tran A, Rey E, d'Athis P, Vincent J, Dulac O, Pons G. Stiripentol in severe myoclonic epilepsy in infancy: a randomised placebo-controlled syndrome-dedicated trial. STICLO study group. Lancet. 2000 Nov 11;356(9242):1638-42. doi: 10.1016/s0140-6736(00)03157-3. PMID 11089822
- [Background] Inoue Y, Ohtsuka Y, Oguni H, Tohyama J, Baba H, Fukushima K, Ohtani H, Takahashi Y, Ikeda S. Stiripentol open study in Japanese patients with Dravet syndrome. Epilepsia. 2009 Nov;50(11):2362-8. doi: 10.1111/j.1528-1167.2009.02179.x. Epub 2009 Jun 22. PMID 19552653
- [Background] Motte J, Trevathan E, Arvidsson JF, Barrera MN, Mullens EL, Manasco P. Lamotrigine for generalized seizures associated with the Lennox-Gastaut syndrome. Lamictal Lennox-Gastaut Study Group. N Engl J Med. 1997 Dec 18;337(25):1807-12. doi: 10.1056/NEJM199712183372504. PMID 9400037
- [Background] Neels HM, Sierens AC, Naelaerts K, Scharpe SL, Hatfield GM, Lambert WE. Therapeutic drug monitoring of old and newer anti-epileptic drugs. Clin Chem Lab Med. 2004;42(11):1228-55. doi: 10.1515/CCLM.2004.245. PMID 15576287
- [Background] Brogden RN, Heel RC, Speight TM, Avery GS. Clobazam: a review of its pharmacological properties and therapeutic use in anxiety. Drugs. 1980 Sep;20(3):161-78. doi: 10.2165/00003495-198020030-00001. PMID 6107238
- [Background] Greenblatt DJ, Divoll M, Puri SK, Ho I, Zinny MA, Shader RI. Clobazam kinetics in the elderly. Br J Clin Pharmacol. 1981 Nov;12(5):631-6. doi: 10.1111/j.1365-2125.1981.tb01281.x. PMID 6120710
- [Background] Giraud C, Tran A, Rey E, Vincent J, Treluyer JM, Pons G. In vitro characterization of clobazam metabolism by recombinant cytochrome P450 enzymes: importance of CYP2C19. Drug Metab Dispos. 2004 Nov;32(11):1279-86. PMID 15483195
- [Background] Jawad S, Richens A, Oxley J. Single dose pharmacokinetic study of clobazam in normal volunteers and epileptic patients. Br J Clin Pharmacol. 1984 Dec;18(6):873-7. doi: 10.1111/j.1365-2125.1984.tb02558.x. PMID 6529527
- [Background] Giraud C, Treluyer JM, Rey E, Chiron C, Vincent J, Pons G, Tran A. In vitro and in vivo inhibitory effect of stiripentol on clobazam metabolism. Drug Metab Dispos. 2006 Apr;34(4):608-11. doi: 10.1124/dmd.105.007237. Epub 2006 Jan 13. PMID 16415114
- [Background] Contin M, Riva R, Albani F, Baruzzi AA. Effect of felbamate on clobazam and its metabolite kinetics in patients with epilepsy. Ther Drug Monit. 1999 Dec;21(6):604-8. doi: 10.1097/00007691-199912000-00004. PMID 10604819
- [Background] Backman JT, Olkkola KT, Aranko K, Himberg JJ, Neuvonen PJ. Dose of midazolam should be reduced during diltiazem and verapamil treatments. Br J Clin Pharmacol. 1994 Mar;37(3):221-5. doi: 10.1111/j.1365-2125.1994.tb04266.x. PMID 8198928
- [Background] Fleishaker JC, Sisson TA, Carel BJ, Azie NE. Pharmacokinetic interaction between verapamil and almotriptan in healthy volunteers. Clin Pharmacol Ther. 2000 May;67(5):498-503. doi: 10.1067/mcp.2000.106292. PMID 10824628
- [Background] Kantola T, Kivisto KT, Neuvonen PJ. Erythromycin and verapamil considerably increase serum simvastatin and simvastatin acid concentrations. Clin Pharmacol Ther. 1998 Aug;64(2):177-82. doi: 10.1016/S0009-9236(98)90151-5. PMID 9728898
- [Background] Lamberg TS, Kivisto KT, Neuvonen PJ. Effects of verapamil and diltiazem on the pharmacokinetics and pharmacodynamics of buspirone. Clin Pharmacol Ther. 1998 Jun;63(6):640-5. doi: 10.1016/S0009-9236(98)90087-X. PMID 9663178
- [Background] Renton KW. Inhibition of hepatic microsomal drug metabolism by the calcium channel blockers diltiazem and verapamil. Biochem Pharmacol. 1985 Jul 15;34(14):2549-53. doi: 10.1016/0006-2952(85)90541-6. PMID 4015695
- [Background] Wang YH, Jones DR, Hall SD. Prediction of cytochrome P450 3A inhibition by verapamil enantiomers and their metabolites. Drug Metab Dispos. 2004 Feb;32(2):259-66. doi: 10.1124/dmd.32.2.259. PMID 14744949
- [Background] Edwards DJ, Lavoie R, Beckman H, Blevins R, Rubenfire M. The effect of coadministration of verapamil on the pharmacokinetics and metabolism of quinidine. Clin Pharmacol Ther. 1987 Jan;41(1):68-73. doi: 10.1038/clpt.1987.11. PMID 3802708
- [Background] Abernethy DR, Egan JM, Dickinson TH, Carrum G. Substrate-selective inhibition by verapamil and diltiazem: differential disposition of antipyrine and theophylline in humans. J Pharmacol Exp Ther. 1988 Mar;244(3):994-9. PMID 3252045
- [Background] Sirmans SM, Pieper JA, Lalonde RL, Smith DG, Self TH. Effect of calcium channel blockers on theophylline disposition. Clin Pharmacol Ther. 1988 Jul;44(1):29-34. doi: 10.1038/clpt.1988.108. PMID 3391002
- [Background] Stringer KA, Mallet J, Clarke M, Lindenfeld JA. The effect of three different oral doses of verapamil on the disposition of theophylline. Eur J Clin Pharmacol. 1992;43(1):35-8. doi: 10.1007/BF02280751. PMID 1505606
- [Background] Allen LV Jr, Erickson MA 3rd. Stability of labetalol hydrochloride, metoprolol tartrate, verapamil hydrochloride, and spironolactone with hydrochlorothiazide in extemporaneously compounded oral liquids. Am J Health Syst Pharm. 1996 Oct 1;53(19):2304-9. doi: 10.1093/ajhp/53.19.2304. PMID 8893069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was recruited from the principal investigator's medical clinic. The other participant contacted us through clincialtrials.gov to participate in this study, and was subsequently recruited because he fit all inclusion/exclusion criteria.
Groups:
- Adjunctive Verapamil: Participants taking verapamil for Dravet syndrome
Period: Overall Study
Arm/Group | Adjunctive Verapamil
Started | 2
Completed | 1
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Open Label Adjunctive Add on: open label adjunctive add on of verapamil to existing medications. dosing begins at 1 mg/kg/d and increases weekly to target of 4 mg/kg/d in divided doses (three times/day)
  Verapamil: Verapamil will be prepared as a solution. A 50mg/ml oral suspension may be made with immediate release tablets and either a 1:1 mixture of Ora-Sweet and Ora-Plus or a 1:1 mixture of Ora-Sweet SF and Ora-Plus will be used.
  Children will start on a 4 weeks titration period:
  Week 1: 1mg/kg/day divided BID Week 2: 2mg/kg/day divided BID or TID Week 3: 3mg/kg/day divided BID or TID Week 4: 4mg/kg/day divided TID
  In event of adverse events, and in consultation with the family and treating physician, the dosage may be decreased to 2mg/kg/day and remain at that dose for the remainder of the study.
Arm/Group | Open Label Adjunctive Add on
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Number of General Tonic-clonic Seizures From Week 8 (Baseline) Visit to Week 12 Visit
Description: The primary study endpoint is the change in number of seizures from baseline. Since we only had one participant finish the study, the endpoint was changed to Week 12 visit. Participants were on verapamil for 4 weeks at Week 12.
Time Frame: Week 8 (baseline) to Week 12
Population: Change in number of general tonic-clonic seizures between Week 8 (baseline) and Week 12 visits.
Measure: Number; unit: General tonic-clonic seizures
Groups:
- Week 8 Baseline: Week 8 visit - 8 weeks of baseline seizure data collected
- Week 12 Verapamil 4mg/kg/Day: Participants have titrated up to 4mg/kg/day of verapamil
Arm/Group | Week 8 Baseline | Week 12 Verapamil 4mg/kg/Day
Number analyzed (Participants) | 2 | 2
General tonic-clonic seizures | 39 | 14

2. Secondary Outcome: Change in Number of Myoclonic Seizures From Week 8 (Baseline) to Week 12
Description: The secondary outcome is the change in number of myoclonic seizures between baseline Week 8 visit and Week 12 visit.
Time Frame: Week 8 (baseline) to Week 12
Population: Participant's collected number of myoclonic seizures at Week 8 visit (baseline) prior to taking verapamil and at Week 12 after 4 weeks of taking verapamil. This participant was the only participant who had seizure types other than general tonic-clonic seizures.
Measure: Number; unit: Myoclonic seizures
Groups:
- Week 8 Baseline: Collected number of seizures at baseline before participants were taking verapamil.
- Week 12 Verapamil 4mg/kg/Day: Participants taking verapamil for 4 weeks post baseline.
Arm/Group | Week 8 Baseline | Week 12 Verapamil 4mg/kg/Day
Number analyzed (Participants) | 1 | 1
Myoclonic seizures | 116 | 175

3. Secondary Outcome: Change in Number of Absence Seizures From Week 8 (Baseline) to Week 12
Description: The secondary outcome measure is the change in number of absence seizures from Week 8 (Baseline) to Week 12
Time Frame: Week 8 to Week 12
Population: Number of Abscence seizures from Week 8 (baseline) to Week 12 visits.
Measure: Number; unit: Abscence seizures
Arm/Group | Week 8 Baseline | Week 12 Verapamil 4mg/kg/Day
Number analyzed (Participants) | 1 | 1
Abscence seizures | 165 | 101

ADVERSE EVENTS:
Time Frame: Up to 35 weeks
Description: Adverse event data was collected from time of consent to end of study participation.
Arm/Group | Open Label Adjunctive Add on
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Adjunctive Add on (N=2)
Seizure (Nervous system disorders) | 1 (1) — Increased frontal lobe seizures up from 0 from the previous visit 4 weeks earlier.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Adjunctive Add on (N=2)
Insomnia (Nervous system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Drooling (Nervous system disorders) | 1 (1) — Increased drooling associated with seizures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No